CLINICAL TRIAL: NCT01722552
Title: China Adherence Through Technology Study
Acronym: CATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: FHI 360 (Other); Guangxi Center for Disease Control and Prevention (Other Government); Dimagi Inc. (Industry); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lora Sabin, Associate Professor, Boston University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R34DA032423-01A1 (NIH)
Record Dates: First submitted 2012-11-03; First posted 2012-11-07 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Medication Adherence
Keywords: HIV; AIDS; antiretroviral therapy; adherence; China
MeSH Terms: conditions — Medication Adherence; Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- adherence feedback (Experimental): Intervention subjects will receive personalized cell phone reminder messages whenever they fail to take a dose within 30 minutes of dose time (as indicated by lack of a Wisepill opening). They will then participate in monthly interactive counseling sessions using summaries of their previous month's behavior. Patients whose mean adherence in the previous month was <95% will be required to have a counseling session, while those with higher adherence will be given the option to have a counseling session.
  Interventions: Behavioral: adherence feedback
- standard of care (Active Comparator): Control subjects will use the electronic monitoring devices just like the intervention arm, but will receive standard of care. They will not receive personalized cell phone reminder messages whenever they fail to take a dose within 30 minutes of dose time, and they will not have access to the summaries of their previous month's behavior for use in interactive counseling sessions, though they will be encouraged to engage in counseling.
  Interventions: Behavioral: standard of care

INTERVENTIONS:
Behavioral: adherence feedback
  Arms: adherence feedback
Behavioral: standard of care
  Arms: standard of care

SUMMARY:
The CATS project is designed to increase understanding of interventions that are feasible and effective in helping injection drug users (IDU) or other patients at high risk of poor medication adherence who are HIV-positive to maintain a high ART adherence. The study will involve: assessing the feasibility and acceptability of using real-time feedback, a wireless technology-updated adaptation of an approach the investigators found to be feasible and effective in China, to promote ART adherence among Chinese patients, including IDU; generating preliminary effectiveness data of real-time feedback on adherence, CD4 count, and HIV viral load; and identifying the factors that explain how real-time feedback influences intervention success or failure.

The specific aims of the study are:

SA1: Determine the feasibility and acceptability of using real-time feedback, a wireless technology-updated adaptation of an approach we found to be feasible and effective in China, to promote ART adherence among Chinese patients. The investigators will conduct a pilot RCT of the real-time feedback intervention among Chinese patients in order to assess its feasibility and acceptability in this population.

SA2: Generate preliminary effectiveness data of real-time feedback on adherence, CD4 count, and HIV viral load. The RCT will allow the researchers to generate rigorous estimates of effect sizes on these important endpoints.

SA3: Describe the factors that explain how real-time feedback influences intervention success or failure. The investigators will use a quantitative-qualitative mixed-methods research approach to explore how the intervention influences the experience of adherence support in this patient population.

DETAILED DESCRIPTION:
The investigators will implement CATS over 2.5 years by implementing a randomized controlled trial to assess real-time feedback, an intervention that utilizes wireless technology via an electronic pill container device ('Wisepill'), and investigating the mechanisms by which the intervention operates using quantitative and qualitative research methods. 120 patients will be enrolled in a HIV clinic in Nanning, capital of Guangxi province, a border province with high rates of HIV and IDU. Enrolled patients will be randomized to intervention vs. comparison group for the 6-month intervention. The study will follow all patients for an additional 3 months to determine sustainability of intervention impact. In addition to adherence and clinical data, quantitative and qualitative data will be collected using survey instruments, focus groups, and in-depth interviews. Analysis of these data will enable achievement of the specific aims and contribute to the scientific evidence base on effective approaches to promoting ART adherence among IDU and other patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years of age and above, currently on ART or about to begin ART at the Guangxi CDC clinic, deemed at risk for poor adherence either by patients or medical staff, own a cell phone, and provide written consent.

Exclusion Criteria:

* Persons who do not speak Mandarin Chinese or who have mental health issues such that they cannot provide written informed consent will not be allowed to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lora Sabin, PhD, Principal Investigator — Boston University Center for Global Health and Development
Locations (2):
- Boston University Center for Global Health and Development, Boston, Massachusetts, United States
- Guangxi CDC ART Clinic, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No
We have no IPD sharing plan.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited subjects from December 2012-April 2013. They were recruited at the Guangxi Provincial ART clinic in Nanning, China. Patients were eligible if they were receiving or initiating antiretroviral therapy (ART), aged 18 years or above, deemed at risk for poor adherence by clinic staff or patients themselves, and owned a mobile phone.
Pre-assignment Details: After enrollment, each subject was given a Wisepill electronic adherence monitoring container for use with his/her ART medications. Subjects selected one or more ART medications to be monitored within the device. All subjects underwent baseline adherence monitoring using Wisepill for 3 months before randomization.
Groups:
- Adherence Feedback: Intervention subjects will receive personalized cell phone reminder messages whenever they fail to take a dose within 30 minutes of dose time (as indicated by lack of a Wisepill opening). They will then participate in monthly interactive counseling sessions using summaries of their previous month's behavior. Patients whose mean adherence in the previous month was <95% will be required to have a counseling session, while those with higher adherence will be given the option to have a counseling session.
  adherence feedback
Period: Overall Study
Arm/Group | Adherence Feedback
Started | 120 (Number of subjects enrolled)
Completed | 116 (Number of subjects who completed the intervention)
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Intervention arm baseline information
Arm/Group | Adherence Feedback
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 63
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Difference in Proportion of Subjects Who Achieve >/= 95% Adherence
Description: Subjects will participate in the 6-month real-time feedback intervention. Comparison patients will continue to be monitored by Wisepill, but they will remain blinded to the adherence information generated by the Wisepill devices, as will their care providers.
Time Frame: Measured at 6 months after start of intervention
Measure: Count of Participants; unit: Participants
Groups:
- Control: Control subjects will use the electronic monitoring devices just like the intervention arm, but will receive standard of care. They will not receive personalized cell phone reminder messages whenever they fail to take a dose within 30 minutes of dose time, and they will not have access to the summaries of their previous month's behavior for use in interactive counseling sessions, though they will be encouraged to engage in counseling.
Arm/Group | Adherence Feedback | Control
Number analyzed (Participants) | 63 | 56
Participants | 55 | 29

2. Secondary Outcome: Proportion of Subjects Who Achieve >/= 95% Cumulative Adherence Over Entire 6 Months of Intervention Period
Description: as for outcome 1
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Adherence Feedback | Control
Number analyzed (Participants) | 63 | 56
Participants | 52 | 29
Statistical Analysis 1: Comparison: Adherence Feedback vs Control; The primary analysis was by intent to treat (ITT). This included data for all randomized subjects, with post-intervention adherence measured by the last 30 days of available data; adherence over the entire 6-month intervention period was measured using all available post-intervention data. Our sample size was designed to detect a 25 percentage point difference in proportion achieving optimal adherence post-intervention; Test type: Equivalence — The margin for non-equivalence was 25 percentage points; p < 0.05, Chi-squared; Risk Ratio (RR) = 1.59, 95% CI 2-sided [1.21 to 2.1]

ADVERSE EVENTS:
Time Frame: Data collection took place from December 2012 and April 2014.
Arm/Group | Adherence Feedback | Control
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/56
Other Adverse Events (participants affected / at risk) | 0/63 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes